CLINICAL TRIAL: NCT04644835
Title: Study of the Effect of Neoadjuvant Low Energy Shock Wave Therapy on Non-Muscle Invasive Bladder Cancer: A Preliminary Pilot Controlled Clinical Trial
Brief Title: Low Energy Shock Wave Therapy and Non-Muscle Invasive Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elkashef, Assistant Lecturer of Urology, Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LESW-NMIBC
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: NMIBC; LESW; TURBT
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LESW group (Experimental): The shock wave applicator (Dornier AR2, shock wave device, Dornier MedTech 2010, Wessling, Germany) will be gently placed directly on the ultrasound transmission gel over the skin surface of the suprapubic region above the urinary bladder at the site of the papillary lesion (ultrasound guided) and at other five points. Points 1 and 2 will be at the level of transverse crease 2 cm above the pubic bone and 5 cm from each, points 3 and 4 will 2 cm above points 1 and 2, and point 5 will be centered of points 1-4. A total of 2000 pulses at 0.25 mJ/mm2 will be delivered with a frequency of 3 pulses per second. The position of the shock wave applicator will be changed after every 400 pulses.
  Interventions: Device: Low Energy Shock Wave Treatment
- Control group (Sham Comparator): This group of patients will be exposed to the same therapy head, which will also be fitted with a stand-off without energy transmission.
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Low Energy Shock Wave Treatment — The shock wave applicator (Dornier AR2, shock wave device, Dornier MedTech 2010, Wessling, Germany) will be gently placed directly on the ultrasound transmission gel over the skin surface of the suprapubic region above the urinary bladder at the site of the papillary lesion (ultrasound guided) and at other five points. Points 1 and 2 will be at the level of transverse crease 2 cm above the pubic bone and 5 cm from each, points 3 and 4 will 2 cm above points 1 and 2, and point 5 will be centered of points 1-4. A total of 2000 pulses at 0.25 mJ/mm2 will be delivered with a frequency of 3 pulses per second. The position of the shock wave applicator will be changed after every 400 pulses.
  Arms: LESW group
Device: Sham Treatment — The patients will be exposed to the same therapy head, which will also be fitted with a stand-off without energy transmission.
  Arms: Control group

SUMMARY:
The investigators hypothesize that low energy shock wave therapy (LESW) might induce damage to the tumor tissues of non-muscle invasive bladder cancer (NMIBC), so they could be ablated and detached from the surface.

The patients who are suffering from NMIBC will be randomly allocated into two groups: The first group (control group): 25 patients will be exposed to sham treatment before transurethral resection of bladder tumor (TURBT) without using LESW therapy. The second group (LESW group): 25 patients will be exposed to LESW therapy before TURBT.

The apoptotic effect of LESW will be studied via histopathological examination and molecular studies of the resected bladder tissues.

The patients will receive intravesical chemotherapy or BCG immunotherapy and they will be followed up at outpatient clinic for two years by MRI, outpatient cystoscopy and cytology to identify the recurrence and progression rate of NMIBC.

DETAILED DESCRIPTION:
The investigators hypothesize that low energy shock wave therapy (LESW) might induce damage to the tumor tissues of non-muscle invasive bladder cancer (NMIBC), so they could be ablated and detached from the surface.

The patients who are suffering from NMIBC will be randomly allocated into two groups: The first group (control group): 25 patients will be exposed to sham treatment before transurethral resection of bladder tumor (TURBT) without using LESW therapy. The second group (LESW group): 25 patients will be exposed to LESW therapy before TURBT. The shock wave applicator (Dornier AR2, shock wave device, Dornier MedTech 2010, Wessling, Germany) will be gently placed directly on the ultrasound transmission gel over the skin surface of the suprapubic region above the urinary bladder at the site of the papillary lesion (US guided) and at other five points. Points 1 and 2 will be at the level of transverse crease 2 cm above the pubic bone and 5 cm from each, points 3 and 4 will 2 cm above points 1 and 2, and point 5 will be centered of points 1-4. A total of 2000 pulses at 0.25 mJ/mm2 will be delivered with a frequency of 3 pulses per second. The position of the shock wave applicator will be changed after every 400 pulses.

The apoptotic effect of LESW will be studied via histopathological examination for the type of bladder tumor, pathological stage, grade, association of carcinoma in situ and morphological features of apoptosis in terms of compaction of the nuclear chromatin (pyknosis), loss of cellular volume and chromatin condensation on the nuclear envelope (nuclear crescents), Immunohistochemical analysis of anti-caspase-3 antibody and molecular studies of Bax (an apoptotic promotor), BCL-2 and Survivin (apoptotic inhibitors) Relative Gene Expression in the resected bladder tissues.

The patients will receive intravesical chemotherapy or BCG immunotherapy and they will be followed up at outpatient clinic for two years by MRI, outpatient cystoscopy and cytology to identify the recurrence and progression rate of NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≤ T1, de novo, single and small (<3cm) papillary lesions will be included in the study.

Exclusion Criteria:

* Patients with ≥ T2 bladder cancer, evidence of nodal metastasis, associated upper tract urothelial carcinoma, morbidly obese patients, patients with absolute contraindication for shock wave therapy or those who refuse will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-28 (Actual); Primary Completion 2022-11-28 (Estimated); Study Completion 2023-11-28 (Estimated)

PRIMARY OUTCOMES:
Progression survival. | 2 years
Recurrence-free survival. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Shokeir, Study Chair — Urology and Nephrology Center, Mansoura University, Egypt; Ahmed Mosbah, Study Director — Urology and Nephrology Center, Mansoura University, Egypt; Ahmed Elkashef, Principal Investigator — Urology and Nephrology Center, Mansoura University, Egypt
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
There is no current plan for whether to share IPD or not.